CLINICAL TRIAL: NCT00070278
Title: A Phase III Randomized Neoadjuvant Study of Sequential Epirubicin/Cyclophosphamide and Paclitaxel + - Gemcitabine in Poor Risk Early Breast Cancer
Brief Title: Neoadjuvant Epirubicin, Cyclophosphamide, and Paclitaxel With or Without Gemcitabine in Treating Women Who Are Undergoing Surgery for Early Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CRUK-neo-tAnGo; CDR0000331863 (Registry Identifier: PDQ (Physician Data Query)); EU-20316
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Gemcitabine; Paclitaxel; Comparative Genomic Hybridization; Microarray Analysis; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Genetic: comparative genomic hybridization
Genetic: microarray analysis
Genetic: mutation analysis
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cyclophosphamide, paclitaxel, and gemcitabine use different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy before surgery may shrink the tumor so that it can be removed during surgery. It is not yet known which combination chemotherapy regimen is more effective in treating early breast cancer.

PURPOSE: This randomized phase III trial is studying different regimens of combination chemotherapy to compare how well they work in treating women who are undergoing surgery for early invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the complete pathological response rate in women with poor-risk early breast cancer treated with neoadjuvant sequential epirubicin, cyclophosphamide, and paclitaxel with vs without gemcitabine.

Secondary

* Compare the disease-free and overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the effect of these regimens on prognostic factors in these patients.
* Correlate molecular profiles, specific gene mutations, and genomic and gene expression changes with clinical outcome in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the health economics associated with this study.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to estrogen-receptor status (negative vs greater than 10% positive cells), HER-2 status (positive vs negative), tumor size (30-50 mm vs greater than 50 mm), and clinical involvement of axillary nodes (yes vs no). Patients are randomized to 1 of 4 treatment arms.

* Neoadjuvant sequential chemotherapy:

  * Arm I: Patients receive epirubicin IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 4 courses. Patients then receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for 4 courses.
  * Arm II: Patients receive paclitaxel as in arm I followed by epirubicin and cyclophosphamide as in arm I.
  * Arm III: Patients receive epirubicin and cyclophosphamide as in arm I followed by paclitaxel as in arm I and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses.
  * Arm IV: Patients receive paclitaxel as in arm I and gemcitabine as in arm III followed by epirubicin and cyclophosphamide as in arm I.
* Surgery: After completion of neoadjuvant chemotherapy, patients in all arms undergo definitive surgery.

Tumor tissue is removed from a subset of patients during serial biopsies. Molecular and genetic profiling, mutation analysis, and comparative genomic analysis is performed on the tissue samples.

Quality of life is assessed at baseline, after 4 courses of chemotherapy, after the completion of chemotherapy, after surgery, and then every 6 months for 2 years.

Patients are followed every 2 months for 2 years and then every 3 months for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 800 patients (200 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Grade 2 or 3
* Tumor size at least 3 cm by ultrasound
* No evidence of metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Not specified

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Fit to receive study chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Complete pathological response after 4 courses

SECONDARY OUTCOMES:
Survival
Disease-free survival
Effect of prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Helena Earl, MBBS, PhD, FRCP — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England, United Kingdom

REFERENCES:
- [Derived] Ali HR, Dariush A, Provenzano E, Bardwell H, Abraham JE, Iddawela M, Vallier AL, Hiller L, Dunn JA, Bowden SJ, Hickish T, McAdam K, Houston S, Irwin MJ, Pharoah PD, Brenton JD, Walton NA, Earl HM, Caldas C. Computational pathology of pre-treatment biopsies identifies lymphocyte density as a predictor of response to neoadjuvant chemotherapy in breast cancer. Breast Cancer Res. 2016 Feb 16;18(1):21. doi: 10.1186/s13058-016-0682-8. PMID 26882907
- [Derived] Abraham JE, Hiller L, Dorling L, Vallier AL, Dunn J, Bowden S, Ingle S, Jones L, Hardy R, Twelves C, Poole CJ, Pharoah PD, Caldas C, Earl HM. A nested cohort study of 6,248 early breast cancer patients treated in neoadjuvant and adjuvant chemotherapy trials investigating the prognostic value of chemotherapy-related toxicities. BMC Med. 2015 Dec 29;13:306. doi: 10.1186/s12916-015-0547-5. PMID 26715442
- [Derived] Earl HM, Vallier AL, Hiller L, Fenwick N, Young J, Iddawela M, Abraham J, Hughes-Davies L, Gounaris I, McAdam K, Houston S, Hickish T, Skene A, Chan S, Dean S, Ritchie D, Laing R, Harries M, Gallagher C, Wishart G, Dunn J, Provenzano E, Caldas C; Neo-tAnGo Investigators. Effects of the addition of gemcitabine, and paclitaxel-first sequencing, in neoadjuvant sequential epirubicin, cyclophosphamide, and paclitaxel for women with high-risk early breast cancer (Neo-tAnGo): an open-label, 2x2 factorial randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):201-12. doi: 10.1016/S1470-2045(13)70554-0. Epub 2013 Dec 19. PMID 24360787